CLINICAL TRIAL: NCT06263530
Title: Prognostic Significance of Circulating Tumor DNA in Hodgkin Lymphoma
Brief Title: Prognostic Significance of ctDNA in HL
Status: Recruiting | Type: Observational
Sponsor: Interni hematologicka klinika FNKV (Network)
Collaborators: Charles University, Czech Republic (Other); General University Hospital, Prague (Other); University Hospital Olomouc (Other); University Hospital Hradec Kralove (Other); University Hospital, Motol (Other)
Responsible Party: Sponsor
Other Study IDs: NU22-03-00182
Record Dates: First submitted 2023-11-14; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Prognostic Cancer Model
Keywords: Hodgkin lymphoma; circulating tumor DNA; next generation sequencing
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Identification of tumor specific mutation profiles at diagnosis of classical Hodgkin lymphoma Quantitative analysis of ctDNA level during the first-line chemotherapy Identification of tumor specific mutation profiles at relapse of classical Hodgkin lymphoma In vitro functional characterization of identified DNA variants and/or mutations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Standard first line treatment, stages I or II without risk factors: Standard first-line treatment that includes 2 cycles of ABVD (doxorubicin, bleomycin, vinblastine, dacarbazine) and involved site radiotherapy of 20 Gy in early clinical stages I or II without risk factors.
- Patients < 60 years, stages I or II and 1 risk factor: Patients below 60 years in intermediate clinical stages I or II with at least one risk factor are treated with 2 cycles of BEACOPP (bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, prednisone) escalated and 2 cycles of ABVD in PET-4 negative cases. Involved site radiotherapy of 30 Gy is indicated in PET-4 positive patients with intermediate stages after chemotherapy.
- Patients < 60 years, stages III or IV with MMT and/or EN disease: Patients in advanced stages III or IV and patients in stage IIB with massive mediastinal tumor and/or extranodal disease are treated with 4 or 6 cycles of BEACOPP escalated based on PET-2 negativity or positivity.
- Elderly patients ≥ 60 years and 1 risk factor: Elderly patients in intermediate stages are treated with 2 cycles of ABVD and 2 cycles of AVD without bleomycin and involved site radiotherapy of 30 Gy.
- Elderly patients ≥ 60 years, stages III or IV: Elderly patients in advanced stages are treated with 2 cycles of ABVD and 4 cycles of AVD without bleomycin
- Relapsed patients up to 65 years: The treatment for patients in relapse up to the age of 65 years is two cycles of platinum based salvage chemotherapy: cisplatin, cytarabine and dexamethasone (DHAP) or ifosfamide, carboplatin, etoposide (ICE) followed by high- dose chemotherapy and autologous stem cell transplantation (ASCT).

SUMMARY:
Specific somatic mutations using ctDNA will be analyzed in predefined subgroups of cHL (e.g., age <60 and ≥ 60 years, EBV). These mutations will be correlated with response to the treatment in the first line, in the relapse, during brentuximab vedotin and/or nivolumab treatment. Circulating tumor DNA will be correlated with the extent of tumor mass and chemo/radiotherapy.

DETAILED DESCRIPTION:
Samples of plasma from peripheral blood will be taken for investigational ctDNA examination during the specific timepoints: at diagnosis, after 2 cycles of initial chemotherapy, at the end of chemotherapy, 3 months after radiotherapy, at the diagnosis of the first relapse, after salvage chemotherapy before ASCT, 3 months after ASCT, at the diagnosis of second relapse and every 3 months during brentuximab vedotin treatment or during nivolumab treatment until progression. The buccal swab for germline DNA extraction will be performed at the time of enrollment into the study. Samples of peripheral blood for EBV-DNA analysis will be obtained from the EBV-positive cHL patients to measure EBV load at the same time-points as ctDNA. Microdissected HRS cells from fresh frozen biopsies at the diagnosis and at the relapse will be used for tumor cells next generation sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years with newly histologically confirmed classical Hodgkin lymphoma (cHL) will be enrolled
* signing the informed consent

Exclusion Criteria:

* Pacients without signing the informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years with new HL, all patients will undergo standard diagnostic procedures and will be divided based by stages and risk factors. Patients below 60 years will be divided into 3 treatment risk groups and treated according to the standard recommendations explained as well as elderly patients (see study groups). Younger relapsed patients will be treated with salvage platinum-based chemotherapy followed by high-dose chemotherapy and autologous stem cell transplantation (ASCT). Relapses after ASCT in younger patients or after at least two lines of chemotherapy in elderly patients will be treated with brentuximab vedotin (up to 16 cycles) or nivolumab until progression.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of tumor specific mutation profiles at dg. of HL based on ctDNA | 4 years
  Identification of tumor specific mutation profiles at diagnosis of classical Hodgkin:
  1. age at diagnosis < 60 years in comparison to patients with age at diagnosis 60 years and more
  2. EBV negative versus EBV positive cases
  3. correlation with the first line treatment outcome lymphoma based on ctDNA analysis with correlation to clinical and pathological characteristics
Quantitative analysis of ctDNA level during the first-line chemotherapy | 4 years
  Quantitative analysis of ctDNA level during the first-line chemotherapy:
  1. analysis in relation to the type of chemotherapy: BEACOPP escalated vs ABVD
  2. dynamics of ctDNA decline in correlation with treatment response
Identification of tumor specific mutation profiles at relapse of classical HL | 4 years
  Identification of tumor specific mutation profiles at relapse of classical Hodgkin lymphoma:
  1. detection of newly developed mutations in comparison to the initial diagnosis
  2. characteristics of mutations in HL tumors refractory to brentuximab vedotin
  3. characteristics of mutations in HL tumors refractory to nivolumab

SECONDARY OUTCOMES:
In vitro functional characterization of identified DNA variants and/or mutations | 4 years
  In vitro functional characterization of identified DNA variants and/or mutations:
  1. variants with unknown impact on classical HL development
  2. variants identified as associated with features analyzed in above mentioned goals

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Mocikova, M.D., Ph.D., Study Chair — Faculty Hospital Kralovske Vinohrady
Locations (5):
- Czechia (5):
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital Kralovske Vinohrady, Prague
  - Charles University, Prague
  - General University Hospital, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dusek L, Majek O. Editorial. Klin Onkol. 2014;27 Suppl 2:3. No abstract available. PMID 25629123
- [Background] Mocikova H, Sykorova A, Stepankova P, Markova J, Michalka J, Kral Z, Buresova L, Belada D. [Treatment and prognosis of relapsed or refractory Hodgkin lymphoma patients ineligible for stem cell transplantation]. Klin Onkol. 2014;27(6):424-8. doi: 10.14735/amko2014424. Czech. PMID 25493581
- [Background] Sykorova A, Mocikova H, Lukasova M, Koren J, Stepankova P, Prochazka V, Belada D, Klaskova K, Gaherova L, Chroust K, Buresova L, Markova J; Czech Hodgkin's Lymphoma Study Group. Outcome of elderly patients with classical Hodgkin's lymphoma. Leuk Res. 2020 Mar;90:106311. doi: 10.1016/j.leukres.2020.106311. Epub 2020 Jan 24. PMID 32050133

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT06263530/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT06263530/ICF_001.pdf